CLINICAL TRIAL: NCT04622618
Title: Optimal Dosing of Preoperative Gabapentin for Prevention of Postoperative Nausea and Vomiting After Abdominal Laparoscopic Surgery: a Randomized Prospective Comparative Study
Brief Title: Optimal Dosing of Preoperative Gabapentin for Prevention of Postoperative Nausea and Vomiting
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Nabil Abdelrahman, Lecturer of anesthesia, Intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FAMSU R 53/2020
Record Dates: First submitted 2020-10-02; First posted 2020-11-10 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Nausea, Postoperative; Vomiting, Postoperative; Pain, Postoperative
Keywords: gabapentin; postoperative nausea and vomiting; laparoscopic surgeries; Visual analogue scale
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: A total of (150) adult patients who will undergo elective abdominal laparoscopic surgery will be included in the study. Written informed consent will be obtained from all patients before randomization. Patients will be divided randomly and equally into three groups (50 patients each(.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Drug formulation will be done by one of the researchers making the dosage of the three groups the same in number and shape of the capsules and then given to a junior anesthetist who is neither involved nor interested in any way in the sample to be administered to the patients surveyed. Blind grouping will be kept to all including the patients themselves, until the completion of the study. Data collection will be done by another anesthesiologist who is blinded to the given medication during the study and not included in the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- G 300 (Active Comparator): The patients will receive 300 mg gabapentin orally 1 hour before induction of anesthesia by a sip of water
  Interventions: Drug: Gabapentin
- G 600 (Active Comparator): The patients will receive 600 mg gabapentin orally 1 hour before induction of anesthesia by a sip of water
  Interventions: Drug: Gabapentin
- G 900 (Active Comparator): The patients will receive 900 mg gabapentin orally 1 hour before induction of anesthesia by a sip of water
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Anticonvulsant, Antiemetic, Analgesic

SUMMARY:
Overall incidence of postoperative nausea and vomiting (PONV) after general anesthesia is 40-90 % . gabapentin has been incorporated into "fast-track" packages and improved recovery during surgery protocols to avoid unintended side effects associated with opioid alternatives. Interestingly, gabapentin has also been noted to reduce the effects of chemotherapy-induced nausea, effective in treatment of gravidarum hyperemesis, and postdural puncture emesis. Different dosing regimens were tested.The goal of the study is to determine the most effective dose of oral gabapentin given 1 hour prior to surgery on the occurrence and severity of PONV and drug side effects in the first 24 hours postoperatively to find the most effective dose of gabapentin with the least side effects.

DETAILED DESCRIPTION:
A total of (150) adult patients who will undergo elective abdominal laparoscopic surgery will be included in the study. Written informed consent will be obtained from all patients before randomization. Randomization will be done with the help of a computer generated list of numbers. Patients will be divided randomly and equally into three groups (50 patients each(. The first group of patients will receive 300 mg gabapentin orally 1 hour before induction of anesthesia by a sip of water (group G1), the second group of patients will receive 600 mg gabapentin orally 1 hour before induction of anesthesia by a sip of water (group G2), the third group of patients will receive 900 mg gabapentin orally 1 hour before induction of anesthesia by a sip of water (group G3). Drug formulation will be done by one of the researchers making the dosage of the three groups the same in number and shape of the capsules and then given to a junior anesthetist who is neither involved nor interested in any way in the sample to be administered to the patients surveyed

ELIGIBILITY:
Inclusion Criteria:

* age between (18- 65) years
* ASA I-II
* scheduled for elective laparoscopic abdominal surgery.

Exclusion Criteria:

* age below 18 and above 60 years
* ASA III- IV
* pregnancy or breastfeeding
* psychiatric illness
* administration of antiemetic or systemic corticosteroids within 24 hours prior to surgery
* vomiting within 24 hours prior to surgery
* alcohol or drug abuse;
* known hypersensitivity or contraindications to gabapentin
* impaired liver or kidney function
* history of motion sickness
* patients on anti-depressants
* patients on whom laparoscopic procedure converted into open technique.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV episodes (nausea, retching or vomiting) | at H4 (4th hour) postoperative
  number of attacks
Incidence of PONV episodes (nausea, retching or vomiting) | at H12 (12th hour) postoperative
  number of attacks
Incidence of PONV episodes (nausea, retching or vomiting) | at H24 (24th hour) postoperative
  number of attacks
Severity of nausea | at H4 (4th hour) postoperative
  measured by nausea verbal numerical rating scale (NVRS) which is an eleven points scale describing nausea severity (0= no nausea, 10= worst nausea imaginable, mild nausea 1-3, moderate 4-6, or severe 7-10)
Severity of nausea | at H12 (12th hour) postoperative
  measured by nausea verbal numerical rating scale (NVRS) which is an eleven points scale describing nausea severity (0= no nausea, 10= worst nausea imaginable, mild nausea 1-3, moderate 4-6, or severe 7-10)
Severity of nausea | at H24 (24th hour) postoperative
  measured by nausea verbal numerical rating scale (NVRS) which is an eleven points scale describing nausea severity (0= no nausea, 10= worst nausea imaginable, mild nausea 1-3, moderate 4-6, or severe 7-10)

SECONDARY OUTCOMES:
Need for rescue antiemetic | during the first 24 hours postoperative
  if severe nausea or two or more emetic episodes, or upon a request from the patient to be repeated if no response within 1 hour up to 3 mg.
Intensity of postoperative pain: Visual Analogue Scale | Total dose in (mg) given during the first 24 hours postoperative
  assessed by using an 11-points Visual Analogue Scale from 0-10 (0= no pain, 10 = worst intolerable pain, mild pain 1-3, moderate pain 4-6, or severe pain 7-10)
incidence of side effects | during the first 24 hours postoperative
  dizziness, headache and somnolence

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - AinShams University, Faculty of medicine, Cairo, Abbasia
  - AinShams University, Faculty of medicine, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Excel sheets of the study
Supporting Information: Study Protocol, SAP
Time Frame: 12 months
Access Criteria: editors of the journal to be submitted to or the corresponding author
URL: http://gharabawy76@yahoo.com